CLINICAL TRIAL: NCT02200289
Title: In Utero Biomass Smoke Exposure, Pro-oxidant/Antioxidant Imbalance and Lung Function in Rural Ghana
Brief Title: In Utero Household Air Pollution Exposure and Lung Development in Ghana
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Columbia University (Other); Kintampo Health Research Centre, Ghana (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1215
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Oxidant Imbalance; Pulmonary Function
Keywords: Birth cohort; Ghana; Biomass; Cook stove; Oxidative stress; Lung development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cord blood, placenta
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mother-infant pairs: Mother-infant pairs from the GRAPHS birth cohort study

SUMMARY:
Household air pollution from cook stoves using solid fuels dominates total population air pollution exposures. Females and young children are disproportionately affected as they either perform or are present for the majority of cooking activities. Worldwide, household air pollution is responsible for 1.6 million premature deaths annually, largely secondary to respiratory tract infections, and 2.7% of worldwide disability-adjusted life years. Children that survive childhood are not free from disease; the WHO estimates that 35% of COPD cases worldwide are secondary to household air pollution. Reducing female and infant morbidity and mortality related to household air pollution secondary to biomass smoke exposure is a top-priority public health goal.

We hypothesize that in utero biomass smoke exposure results in a fetal oxidant imbalance, which negatively impacts lung development. We will leverage the success of the Ghana Randomized Air Pollution and Health Study, a randomized cook stove intervention trial of 1,415 mother-infant pairs, to examine the impact of maternal household air pollution exposure on cord blood oxidant imbalance and infant pulmonary function. We aim to enroll at least 150 infants, analyze cord blood samples for markers of oxidant imbalance and perform infant pulmonary function testing. Cord blood will also be prepared for future immune, hormonal and epigenetic testing. This study will allow us to consider interventions, such as maternal antioxidant dietary supplementation during pregnancy, to compliment existing cook stove interventions and reduce household air pollution-related morbidity and mortality.

DETAILED DESCRIPTION:
The proposed study will be nested within the Ghana Randomized Air Pollution and Health Study (GRAPHS) to investigate oxidant imbalance and pulmonary function in infants exposed to in utero household air pollution.

GRAPHS is a birth cohort study examining the impact of reduced maternal household air pollution exposure on birth outcomes and incident infant pneumonia. Mother-infant pairs are recruited from the Kintampo Health Research Centre (KHRC) catchment area in rural Ghana, which comprises a population of 146,000 people. 1,415 nonsmoking women who primarily deliver at one of four KHRC birth facilities and are pregnant with a singleton fetus of gestational age less than 24 weeks are eligible for participation. After enrollment, women are randomized to a no-emission liquid petroleum gas (LPG) stove, a low-emission BioLite cook stove or control (high-emission) arms and undergo four 72-hour carbon monoxide (CO) and/or particulate matter (PM) prenatal exposure monitoring sessions. Birth weights and outcomes are recorded and a placenta sample is stored in formalin for future analyses. The infants are followed with CO and PM exposure monitoring sessions at 1, 3 and 9 months of age and weekly surveillance for incident respiratory disease.

For the proposed study, we will recruit and consent GRAPHS mother-infant pairs. Venous cord blood and placenta samples will be collected following placenta delivery. Cord blood will be placed on IsoRack cool packs designed to maintain samples at 0°C for up to 6 hours. Cord blood samples will be processed for biomarkers of oxidant imbalance and for future study, including but not limited to immune function, hormonal balance and epigenetic analyses. After initial processing, samples will be frozen at -80°C until oxidant analyses are performed using commercially available reagent kits and protocols.

When the infant is one month old or younger, trained study personnel will perform noninvasive pulmonary function testing (PFT) using the Medispirit Whistler Lung Function Measurement Instrument (LFMI) in accordance with ATS/ERS guidelines. The Medispirit Whistler LFMI is a lightweight and portable device that allows non-invasive PFTs to be performed in the infant's home. The Whistler LFMI flow measurement is ultrasonic and therefore does not need to be calibrated. The infant will be held with his/her head in a stable position until s/he is breathing quietly or asleep. A sterile, single-use, transparent facemask that does not interfere with normal breathing will be placed over the infant's mouth and nose. Tidal flow volume loops will be recorded and single occlusion test will be used to determine the ratio of time to reach peak expiratory flow to total expiratory time, compliance and resistance.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Primarily deliver at one of four KHRC birth facilities
* Pregnant with a singleton fetus
* Pregnancy of gestational age less than 24 weeks

Exclusion Criteria:

* Pregnant with more than a singleton fetus (twins, etc)
* Pregnancy beyond 24 weeks gestation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mother-infant pairs are recruited from the Ghana Randomized Air Pollution and Health Study (GRAPHS). GRAPHS participants are from the Kintampo Health Research catchment area in rural Ghana, which comprises a population of 146,000 people.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Oxidant imbalance | Day 1
  at infant delivery

SECONDARY OUTCOMES:
Lung function | up to 1 month
  Infant age less than or equal to one month

CONTACTS AND LOCATIONS:
Overall Officials: Alison Lee, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Kintampo Health Research Centre, Kintampo, Ghana